CLINICAL TRIAL: NCT06739525
Title: The Effects of Blue of Blue Light-blocking Glasses Versus Standard Lenses on Contrast Sensitivity & Visual Fatigue in Myopic & Non-Myopic Adults
Brief Title: Effects of Blue of Glasses VS Standard Lenses on Contrast Sensitivity & Visual Fatigue in Myopic & Non-Myopic Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/749
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental)
  Interventions: Combination Product: Blue Light-Blocking Glasses (Intervention Group)
- Control Group (Active Comparator)
  Interventions: Diagnostic Test: Standard Lenses (Control Group)

INTERVENTIONS:
Combination Product: Blue Light-Blocking Glasses (Intervention Group) — Participants in this arm wore blue light-blocking glasses designed to filter out a portion of short-wavelength blue light. These lenses were intended to reduce eye strain and protect against blue light exposure, especially during prolonged screen time. Participants used blue light-blocking glasses consistently throughout the study period to assess their effect on contrast sensitivity and visual fatigue.
  Arms: interventional group
Diagnostic Test: Standard Lenses (Control Group) — Participants in this arm wore standard lenses without any blue light-blocking properties. These lenses allow the full spectrum of visible light to pass through and serve as a baseline control to measure against the blue light-blocking glasses. Participants used these lenses under the same conditions to assess contrast sensitivity and visual fatigue without blue light filtration.
  Arms: Control Group

SUMMARY:
This study investigates the effects of blue light-blocking glasses compared to standard lenses on contrast sensitivity and visual fatigue in myopic and non-myopic adults. With the growing use of digital screens, blue light exposure has raised concerns due to potential eye strain, sleep disruption, and visual fatigue.

DETAILED DESCRIPTION:
While blue light-blocking lenses are marketed to address these issues, evidence of their efficacy, particularly for different refractive errors like myopia, remains inconclusive. Using a randomized controlled design, this study will assess both groups across specific visual tasks to measure contrast sensitivity and visual fatigue. Outcomes are evaluated using validated tools, including the Computer Vision Syndrome Questionnaire (CVS-Q) and Visual Fatigue Questionnaire (VFQ), with measurements taken at baseline, 2 weeks, and 4 weeks. Findings are expected to clarify the potential advantages of blue light-blocking glasses over standard lenses, aiding in evidence-based recommendations for adults with varying visual needs.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-50 years.
* Both myopic (with any degree of myopia) and non-myopic adults.
* Participants who use computer screens for at least four hours per day.
* Individuals currently using corrective lenses or willing to wear study-provided glasses during the experiment.
* Individuals willing to complete the study protocol, which includes attending follow-up examinations and filling out visual fatigue questionnaires.

Exclusion Criteria:

* A history of any serious vision-related condition (such as glaucoma, cataracts, or retinal problems).
* Individuals who have already undergone refractive surgery (e.g., LASIK) or other types of eye surgery.
* Systemic conditions affecting vision include diabetes, neurological problems, and any other ailment that may impair visual ability.
* Taking drugs that are known to impair vision or produce visual tiredness (for example, certain antihistamines and antidepressants).
* Pregnant women's visual performance may be affected by hormonal changes.
* People with uncorrected vision difficulties cannot use the prescription lenses during study time.
* Participants who are allergic or sensitive to lens materials.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Contrast Sensitivity | 12 Months
  Measured using the Pelli-Robson chart to assess changes in visual acuity and sensitivity to contrast under different lens conditions.
Visual Fatigue | 12 months
  The Visual Fatigue Questionnaire (VFQ) was assessed to evaluate subjective experiences of eye strain and fatigue during visual tasks.
  Computer Vision Syndrome: Evaluated with the Computer Vision Syndrome Questionnaire (CVS-Q) to quantify symptoms associated with prolonged screen use, including dryness, discomfort, and eye strain."

CONTACTS AND LOCATIONS:
Locations (1):
- Tehsil Headquarters (THQ), Taunsa, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No